CLINICAL TRIAL: NCT03187041
Title: Skin Surface Pressures Under Blood-Draw Tourniquets
Brief Title: Sensation and Skin Pressures Under Blood-Draw Tourniquets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 161885
Record Dates: First submitted 2017-06-09; First posted 2017-06-14 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Skin Pressures Under Blood Draw-tourniquets
Keywords: blood draw tourniquets; skin surface pressure; blood draw band; elastic tourniquet; phlebotomy; tourniquet pressure
MeSH Terms: interventions — Sensation

STUDY DESIGN:
Intervention Model Description: In order to acquire our data, a Microlab PicoPress device will be employed. It has been shown to provide accurate, linear, and reproducible measures of surface pressure between the skin and device. For tourniquets, the investigators will be using a MedSource perforated tourniquet, which is the type of elastic tourniquet the phlebotomists are accustomed to using in their daily practice. For each experiment throughout both phases of the study, the PicoPress pressure sensor will be folded in half and taped over the lateral aspect of the right arm, approximately 2 inches distal to the deltoid muscle along the brachialis muscle. Arm circumferences will be taken prior to experimentation at this same location. For each trial, the phlebotomists will tie the 2.5cm elastic tourniquet around the arm and pressure sensor while ensuring that the tourniquet is not knotted directly on top of the sensor. The study will be divided into two phases of experimentation conducted sequentially.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Skin surface pressures under tourniquets and sensation (Experimental): Phase 1: Each phlebotomist will apply the tourniquet 10 separate times to the right arm of each subject. The tourniquet will remain on the arm for approximately ten seconds, to be able to allot enough time to collect an accurate pressure measurement. All 10 tourniquet skin pressure measurements will take place on the same day for a subject.
  Phase 2: 20 subjects will be subjected to a prolonged blood-draw tourniquet application for a duration of 1 hour. The purpose of phase 2 is to determine whether there is an effect on sensation from prolonged blood tourniquet use.
  Interventions: Other: Sensation and Skin Surface Pressures Under Blood-Draw Tourniquets

INTERVENTIONS:
Other: Sensation and Skin Surface Pressures Under Blood-Draw Tourniquets — Phase 1: Skin surface pressures will be recorded by an investigator during each of the 10 applications of the tourniquet. All 10 tourniquet skin pressure measurements will take place in the Blood Draw clinic at the UCSD Medical Center in Hillcrest on the same day for a subject.
  Phase 2: The same 20 subjects will be subjected to a prolonged blood-draw tourniquet application for a duration of 70 minutes. The purpose of phase 2 is to determine whether there is an effect on sensation from prolonged blood tourniquet use. External skin pressures will not exceed 60mmHg. During this prolonged tourniquet application the investigators will monitor changes in hand sensation at 10-minute intervals using Semmes-Weinstein monofilaments on three peripheral nerves of the hand (median, radian, and ulnar).

SUMMARY:
Purpose: This research study seeks to determine whether surface pressures generated by elastic tourniquets used by phlebotomists during blood-draws can penetrate to deeper tissues where major arteries and nerves lie. Additionally, investigators will also determine the effects of prolonged tourniquet application on hand sensation using a controlled, reproducible force stimulus. In conjunction, the investigators will also track changes in skin surface pressures and pain levels over this prolonged tourniquet application. Hypothesis: The investigators hypothesize the use of common elastic tourniquets used for blood draws does not significantly impact sensation and will not elicit nerve or tissue damage. Technologies used: Monofilaments and Pressure Sensor

DETAILED DESCRIPTION:
The objective of this study is to investigate the reproducibility and consequently the safety of common elastic tourniquet methods for blood draws. Specifically, the study will investigate whether the surface pressures produced by blood draw tourniquets when applied by experienced phlebotomists are significant enough to penetrate to deeper tissue near bone where major arteries and nerves lie. By relating factors including tourniquet width and patient arm circumference to our surface pressure measurements and comparing our results to previous literature, the investigators hope to determine the safety of current blood draw tourniquet procedures.

In addition, the investigators will track changes in skin surface pressures over time to determine if prolonged exposure to these tourniquet pressures has the potential to permanently affect nerve function and muscle in tissues near bone.

Hand sensation will be investigated during a prolonged tourniquet application trial of the study to test the effects of the generated pressures on median, ulnar, and radial nerve viability over time.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older

Exclusion Criteria:

* no history of abnormal heart conditions
* no history of coagulation disorders
* will not be on prescription medications that affect cardiovascular system (ex: medications that affect blood pressure or cardiac contractility etc.)**
* does not have diabetes

  * Types of medications that affect the cardiovascular system and are part of the exclusion criteria include but are not limited to: anticoagulants, antiaginals, antiarrhythmic agents, anti-hypertensive/hypotensive agents, cardenolides, cardiac stimulants, hypolipidemic agents, inotropic agents, vasoconstrictors, as well as vasodilators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Skin Surface Pressure Under Blood-Draw Tourniquet with Phlebotomists (Phase 1) | Phase 1: 10-15 seconds (10 times within a 5 -10 minute period)
  The pressure under blood draw tourniquets will be taken in Phases 1 and 2. During phase 1, the tourniquet will remain on the subject for a brief period of time (10-15 seconds) 10 times, allowing for enough time to acquire pressure measurements using the PicoPress device. The difference between Phase 1 and Phase 2 is that phase 1 will be performed with a phlebotomist, while phase 2 will be performed with one of the investigators for an extended period of time.
Skin Surface Pressure Under Blood-Draw Tourniquet and Change in sensation during a 1 hour period (Phase 2) | Phase 2: 70 minutes (sensation will be measured every 10 minutes)
  Phase 2: The PicoPress will constantly monitor pressure under the arm tourniquet for one hour. The investigators will also simultaneously monitor the changes from baseline in sensation using Semmes-Weinstein Monofilaments on the radial, ulnar, and median nerves in participants.

CONTACTS AND LOCATIONS:
Overall Officials: Alan R Hargens, PhD, Principal Investigator — UCSD
Locations (1):
- UC San Diego Medical Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared.

REFERENCES:
- [Background] Crenshaw AG, Hargens AR, Gershuni DH, Rydevik B. Wide tourniquet cuffs more effective at lower inflation pressures. Acta Orthop Scand. 1988 Aug;59(4):447-51. doi: 10.3109/17453678809149401. PMID 3421083
- [Background] Partsch H, Mosti G. Comparison of three portable instruments to measure compression pressure. Int Angiol. 2010 Oct;29(5):426-30. PMID 20924346